CLINICAL TRIAL: NCT03833765
Title: Adjunctive Benefit of a Xenogenic Collagen Matrix Associated With Coronally Advanced Flap for Treating Multiple Gingival Recessions
Brief Title: Adjunctive Benefit of a Xenogenic Collagen Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roberto Rotundo (Individual)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Roberto Rotundo, Principal Investigator, Rotundo, Roberto, DDS
Organization: Rotundo, Roberto, DDS (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STXen
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Gingival Recession
Keywords: gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: single-centre, superiority, double blind clinical trial, with balanced randomisation and parallel two groups design according to CONSORT statement
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAF+XCM (Experimental): An envelope split-full-split thickness flap without vertical incisions will be carried out in the gingival recession area. Afterwards, a xenogenic collagen matrix (XCM) will be applied to all teeth with recession defect. The XCM will be cut into the right dimensions, measured with the probe, and its measurements recorded; then it will be placed from the CEJ to the bone crest on the recipient bed using single sutures, 7/0 PGA sutures. The matrix will be rehydrated with blood, in order to reconstitute and maintain the maximal thickness possible. The flap will be closed slightly coronal to the CEJ with a sling suture using resorbable PGA 6/0 sutures and avoiding any compression of the matrix.
  Interventions: Procedure: CAF+XCM
- CAF alone (Active Comparator): An envelope split-full-split thickness flap without vertical incisions will be carried out. The root surfaces will be mechanically treated with the use of curettes. A sharp dissection into the vestibular lining mucosa will be then carried out to eliminate muscle tension. Sling sutures will be performed to accomplish a precise adaptation of the buccal flap on the exposed root surfaces and to stabilize every single surgical papilla over the de-epithelialized anatomic papillae.
  Interventions: Procedure: CAF alone

INTERVENTIONS:
Procedure: CAF+XCM — After flap elevation according to the Coronally Advanced Flap procedure for multiple recession defects, a Xenogeneic Collagen Matrix was applied and then covered by the flap.
  Arms: CAF+XCM
Procedure: CAF alone — Coronally Advanced Flap procedure alone was performed to treat multiple recession defects
  Arms: CAF alone

SUMMARY:
The present CONSORT-based randomized clinical trial is to assess the adjunctive benefit of a xenogenic collagen matrix in combination with a coronal advanced flap with respect to a coronal advanced flap alone in the treatment of multiple gingival recession defects in adult population.

DETAILED DESCRIPTION:
This is a single-centre, superiority, double blind clinical trial, with balanced randomisation and parallel two groups design. The 2 groups will be:

1. CAF combined with XCM;
2. CAF alone.

The objective is therefore to assess the adjunctive benefit of a xenogenic collagen matrix in combination with a coronal advanced flap.

The primary endpoint is the mean recession reduction after 6 and 12 months post treatment.

The secondary endpoints are: Percentage of complete root coverage after 6 and 12 month; Thickness of soft tissue over the root after 6 and 12 month; Recession width after 6 and 12 month; KT width; Patients satisfaction.

The following Inclusion Criteria have to be satisfied: patient (male or female) must be 18 years or older, not pregnant, and candidate for buccal root coverage procedure in the upper jaw; recession defects have to be AAA or ABA (according to Rotundo et al classification), with at least 2 adjacent RC with ≥ 2 mm RC depth and root abrasion depth less than 1 mm; Patient shows sufficient plaque control (FMPS ≤ 20%) and acceptable bleeding score(FMBS ≤ 20%); Teeth intended to treat are in the region 1 - 5; patient has to be able to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures; patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent.

Randomisation: Computer-generated blocked for each centre, with allocation concealment by opaque sequentially numbered sealed envelopes.

Blinding: Patients and outcome assessor blind to group assignment.

Sample size: Based on a formula for cluster design to detect a difference between treatments of 1 mm in recession reduction (standard deviation of 0.93 mm - Woodyard et al. 2004) with a two-side 5% significance level, a power of 90%, a mean number of treated teeth per patient of 2.92, an intraclass correlation coefficient of 0.35, a sample size of 24 patients per treatment will be necessary.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (male or female) must be 18 years or older
2. Presence of gingival recessions in the upper jaw, involving teeth from central incisor to first molar
3. Gingival recessions on at least 2 adjacent teeth with a minimal depth of 2mm and detectable cemento-enamel junction (CEJ) (abrasion step <1mm)
4. The patient is able to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures
5. Full Mouth Plaque (FMPS) and Bleeding (FMBS) Score <20%
6. The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent

Exclusion Criteria:

1. Smoker patients
2. Pregnant patients
3. Patients affect by uncontrolled diabetes
4. General contraindications for dental and/or surgical treatment are present
5. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years
6. The patient is taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs, anticoagulation drugs)
7. The patient has a disease, which affects connective tissue metabolism (e.g. collagenases)
8. The patient is allergic to collagen
9. The patient is an abuser of alcohol or drug
10. Patients have participated in a clinical trial within the last six months
11. Presence of untreated periodontitis
12. Gingival recessions on molar teeth (excluding the first) or on malpositioned teeth
13. Presence of abrasion ≥ 1 mm or cervical restoration, with non-detectable CEJ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Mean Recession Reduction | 12 months
  The distance between CEJ and the free gingival margin (Rec depth) will be measured at baseline, 3, 6 and 12 months. The mean change will be then calculated.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03833765/Prot_SAP_000.pdf